CLINICAL TRIAL: NCT06192355
Title: One-Scope II: Single-use Versus Reusable Gastroscopes in Patients With Upper Gastrointestinal Bleeding.
Brief Title: Single-use Versus Reusable Gastroscopes in Patients With Upper Gastrointestinal Bleeding.
Acronym: OneScopeII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00000013
Record Dates: First submitted 2023-05-12; First posted 2024-01-05 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Endoscopy; Emergency
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-use gastroscope (Experimental): A disposable endoscope designed for a one-time use during a Gastroscopy, eliminating the need for reprocessing or sterilization. After a single procedure, the entire gastroscope is discarded, reducing the risk of cross-contamination and ensuring a fresh, sterile instrument for each patient intervention
  Interventions: Device: Endoscopic hemostasis using a Esophagogastroduodenoscopy
- reusable gastroscope (Active Comparator): A durable endoscope designed for multiple uses after thorough reprocessing and sterilization
  Interventions: Device: Endoscopic hemostasis using a Esophagogastroduodenoscopy

INTERVENTIONS:
Device: Endoscopic hemostasis using a Esophagogastroduodenoscopy — performing an Esophagogastroduodenoscopy for diagnosis and therapy of possible bleeding sites

SUMMARY:
Controlled-randomized trial evaluating single-use versus reusable gastroscopes in patients with upper gastrointestinal bleeding.

DETAILED DESCRIPTION:
Acute upper gastrointestinal bleeding is a common medical emergency. According to guidelines, endoscopic evaluation should be performed within 24 hours. With an overall high incidence and an overall high number of diagnostic and therapeutic endoscopic procedures, the introduction of new endoscopic concepts may have a profound impact on outcomes as well as cost-effectiveness in upper gastrointestinal bleeding. For this purpose, the use of single-use gastroscopes represents an interesting possibility. Hygiene issues in the emergency situation are also relevant. The previous feasibility study One-Scope I demonstrated that the diagnosis as well as the therapy of upper gastrointestinal bleeding is possible with single-use gastroscopes. In this follow-up study, the investigators compare the use of single-use versus reusable gastroscopes in participants with suspected upper gastrointestinal bleeding in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow-Blatchford score (GBS) >2
* Clinical signs of upper bleeding

Exclusion Criteria:

* pregnancy
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
intraprocedural technical success | Up to 20 minutes
  defined as reaching the descending duodenum and adequately assessing for the presence of a bleeding site

SECONDARY OUTCOMES:
intraprocedural clinical success | Up to 45 Minutes
  defined as successful endoscopic hemostasis during the examination if required
re-bleeding rate | Up to 30 days
  need for further endoscopic, interventional-angiographic, or surgical intervention within 30 days due to upper GI-bleeding
blood transfusions | Up to 30 days
  Need for blood transfusion due to a hemorrhage-related decrease in hemoglobin levels ≤ 70 g/L
Length of Stay | Up to 30 days
  Duration of inpatient stay, measured from the day of admission to the day of discharge
Length of intervention | Up to 60 minutes
  measured from initiation to achievement of hemostasis
cross over to reusable gastroscope | Up to 60 Minutes
  Switch to a reusable gastroscope in case of non-achieved technical or clinical success, such as unsuccessful hemostasis, insufficient assessment of the bleeding source, or inability to reach the descending duodenum
Adverse events | Up to 30 days
  Occurrence of adverse events, such as perforation, bleeding exacerbation, aspiration, and infection.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Römmele, MD, Principal Investigator — Unervsity Hospital Augsburg
Locations (1):
- University Hospital of Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No